CLINICAL TRIAL: NCT04185324
Title: Effectiveness of Visual Cues and Verbal Storytelling in Teaching Preschool Children Zippering
Brief Title: Efficacy of an Intervention to Teach Zippering: A Two-Group Control Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SalusU
Record Dates: First submitted 2019-11-26; First posted 2019-12-04 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2019-12

CONDITIONS: Typical Preschoolers Who Can Not Zipper
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: two cohort
Who Masked: Participant, Care Provider
Masking Description: Preschoolers are not aware of whether they receive zippering instruction using a standard teaching zippering vest or the modified one. The parents were not aware which group their child was put in. All children received extra practice with zippering, in both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard zippering vest (Experimental): Children receive three supervised sessions for them to practice engaging and pull up a zipper, using a standard teaching zippering vest.
  Interventions: Behavioral: Standard zippering vest
- Modified zippering vest (Experimental): Children receive three sessions of specially designed zippering instruction using a modified zippering vest, where they can practice engaging and pulling up a zipper after being read a related story.
  Interventions: Behavioral: Modified zippering vest

INTERVENTIONS:
Behavioral: Standard zippering vest — Standard zippering vest used to teach zippering
  Other Names: Control group
  Arms: Standard zippering vest
Behavioral: Modified zippering vest — Modified zippering vest used to teach zippering, along with related story
  Other Names: Comparison group
  Arms: Modified zippering vest

SUMMARY:
Preschoolers are assigned to a control group or a comparison group to examine the efficacy of a new intervention to teach the skill of engaging and pulling up a zipper.

DETAILED DESCRIPTION:
Purpose: This pilot study compares the efficacy of a standard teaching zippering vest presented with general verbal prompts to a modified teaching zippering vest presented with a related story and vocabulary in the acquisition of zippering skills among typically developing preschoolers. Institutional Review Board approval and parent consent was obtained.

Design: An experimental two group pre-post test design was used. Setting: Research occurred in a local preschool. Participants: Participants were recruited from fifty 3.6-to 4.11-year-old preschoolers.

Intervention: Eligible children received 3 zippering practice sessions with either a standard zippering vest (control group) or a modified vest with added visual and language cues (comparison group).

The treatment protocol for both cohorts of participants was administered over a three-week time period to minimize the impact of normal development.

ELIGIBILITY:
Inclusion Criteria: Child must be typically developing as assessed by the Developmental Assessment of Young Children 2 (DAYC-2) developmental screening.

Child must be between 42 and 60 months of age. Child must be unable to zip by a) parent report and b) three observed attempts to zipper -

Exclusion Criteria:

Child must meet inclusion criteria and be present at school during three researcher visits to the preschool within three consecutive weeks.

-

Ages: 42 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Zippering steps completed | all data was collected within three weeks for each child to minimize the impact of typical development
  The task of engaging and pulling up a zipper was broken down to 7 steps. By examining video data, the number of zippering steps completed was analyzed for each zippering trial.

CONTACTS AND LOCATIONS:
Overall Officials: Fern Silverman, EdD, Principal Investigator — Salus University
Locations (1):
- Little Joes preschool, Jenkintown, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No